CLINICAL TRIAL: NCT00408096
Title: Comparison of Two Resurfacing Prostheses in the Treatment of Osteoarthritis of the Shoulder A Prospective, Randomized Migration and Bone Density Study
Brief Title: Comparison of Two Resurfacing Prostheses in the Treatment of Osteoarthritis of the Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20060165
Record Dates: First submitted 2006-12-05; First posted 2006-12-06 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2014-10

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; shoulder; resurfacing; prosthesis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): The Copeland uncemented prostheses with titanium-sprayed, hydroxyapatite (HA)-coated bone-contact area used as a treatment for shoulder osteoarthritis
  Interventions: Procedure: Copeland or Global CAP resurfacing prosthesis
- 2 (Active Comparator): The Global Cap uncemented prostheses with titanium-sprayed, hydroxyapatite (HA)-coated bone-contact area used as a treatment for shoulder osteoarthritis
  Interventions: Procedure: Copeland or Global CAP resurfacing prosthesis

INTERVENTIONS:
Procedure: Copeland or Global CAP resurfacing prosthesis — Both Copeland and Global Cap are uncemented prostheses with titanium-sprayed, hydroxyapatite (HA)-coated bone-contact surfaces.

SUMMARY:
The purpose of this study is to determine whether there is a difference between the result of treatment of shoulder osteoarthritis with two different shoulder prostheses.

DETAILED DESCRIPTION:
In this randomized study, we wish to investigate with the use of clinical and radiological parameters whether there is a difference between the result of treatment of shoulder osteoarthritis with the Copeland resurfacing prosthesis and the Global CAP resurfacing prosthesis.

Clinical parameters with the help of the Constant Shoulder Score (CSS) and Western Ontario Osteoarthritis of the Shoulder Index (WOOS):

1. Pain
2. Activities of Daily Living (ADL)
3. Range of Motion (ROM)
4. Muscle strength

Radiologic parameters:

1. Migration of resurfacing prostheses with use of MB-RSA
2. Bone density around the prosthesis measured with Dual Energy X-ray Absorptiometry (DEXA)
3. Correlation between bone density and prosthesis migration

ELIGIBILITY:
Inclusion Criteria:

1. Patients with shoulder osteoarthritis with cartilage defect of the caput humeri and not the glenoid cavity
2. Aged 18 years or older and fit
3. Informed, written consent -

Exclusion Criteria:

1. Patients found unsuitable preoperatively for a resurfacing prosthesis
2. Patients aged 85 or older
3. Patients with rheumatoid arthritis
4. Patients who previously had undergone shoulder alloplasty or other major shoulder surgery (more than just diagnostic arthroscopy)
5. Patients unable to avoid NSAID after surgery
6. Patients requiring regular systemic steroid treatment
7. Female patients taking hormone substitution
8. Patients with metabolic bone disease
9. Severe shoulder instability with large rotator cuff defect ( will often necessitate special prosthesis components or even major soft-tissue surgery)
10. Female patients in the fertile age range who do not use safe anti-conception (oral contraception, intrauterine devices, depot gestagens, vaginal hormone rings) -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-12; Primary Completion 2016-03 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Migration of resurfacing prostheses | five years
Bone density around the prosthesis | five years
Pain | five years
Activities of Daily Living (ADL) | five years

SECONDARY OUTCOMES:
Range of Motion (ROM) | five years
Muscle strength | five years
Correlation between bone density and prosthesis migration | five years

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Soballe, Professor, Study Director — Orthopaedic Department, Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Orthopaedic Department K, Silkeborg Hospital, Silkeborg
  - Regionshospitalet Viborg, Viborg

REFERENCES:
- [Derived] Jorgensen PB, Krag-Nielsen N, Lindgren L, Morup RMS, Kaptein B, Stilling M. Radiostereometric analysis: comparison of radiation dose and precision in digital and computed radiography. Arch Orthop Trauma Surg. 2023 Sep;143(9):5919-5926. doi: 10.1007/s00402-022-04674-0. Epub 2022 Nov 23. PMID 36422666
- [Derived] Mechlenburg I, Klebe TM, Dossing KV, Amstrup A, Soballe K, Stilling M. Evaluation of periprosthetic bone mineral density and postoperative migration of humeral head resurfacing implants: two-year results of a randomized controlled clinical trial. J Shoulder Elbow Surg. 2014 Oct;23(10):1427-36. doi: 10.1016/j.jse.2014.05.012. PMID 25220196